CLINICAL TRIAL: NCT05100758
Title: Effect of Active Hexose Correlated Compound to Clinical and Immunological Response in Tuberculosis-HIV (Human Immunodeficiency Virus) Infection
Brief Title: Active Hexose Correlated Compound in Tuberculosis-HIV (Human Immunodeficiency Virus) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0307210724
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus
Keywords: Active Hexose Correlated Compound; Tuberculosis-HIV; Cytokine; Sputum Conversion
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: One group will be given Active Hexose Correlated Compound as adjuvant and the comparison group will only receive the tuberculosis treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will be blinded from the allocation (not allowed to observe the allocation and intervention) and the outcome assessor will not be informed the code of allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Hexose Correlated Compound (Experimental): The participants will be given Active Hexose Correlated Compound as a capsule 3 gram/ daily for 6 months
  Interventions: Dietary Supplement: Active Hexoses Correlated Compound
- Control Group (No Intervention): Participant will be given only the tuberculosis and antiretroviral treatment

INTERVENTIONS:
Dietary Supplement: Active Hexoses Correlated Compound — Active Hexose Correlated Compound was isolated from basidiomycetes which comprise polysaccharides and amino acids.
  Arms: Active Hexose Correlated Compound

SUMMARY:
Background

Active Hexose Correlated Compound is assumed to have a positive effect on immunity, including induce a phagocytic response, reduce tumor resistance, and cytokine response including interferon-gamma and interleukins. Tuberculosis patients with concurrent Human immunodeficiency Virus (HIV) might have benefit when receiving active hexose compound during tuberculosis treatment

Purposes

1. To assess the clinical changes of patients who receive active hexose compound as an adjuvant to tuberculosis therapy in patients with HIV
2. To assess the difference of pro-inflammatory cytokines between standard therapy and active hexose compound adjuvant

Methods A clinical trial involving patients with Tuberculosis-HIV infection

Hypothesis

1. Clinical improvement is significantly different where the group who receive active compound will have the better clinical outcome
2. Lower proinflammatory cytokines are observed in people who receive active compound

DETAILED DESCRIPTION:
Population :

Lung Tuberculosis patient with HIV Infection

Design :

Double-Blind Randomized Control Trial at the outpatient setting

Randomization Simple Randomization

Proposed Number of participants :

Using the difference between two independent means of duration to sputum conversion

1. Type 1 error 5%
2. Power of study 80%
3. Effect Size 0.5
4. Dropout rate 20% Total Participant 122

Proposed analysis

1. Time-to-event analysis using cox regression for the duration of sputum conversion and radiology resolution
2. Linear mixed model for continuous dependent variable

ELIGIBILITY:
Inclusion Criteria:

1. Newly-diagnosed Lung Tuberculosis case who will receive a 6-month regiment
2. Not Pregnant
3. Diagnosed with HIV

Exclusion Criteria:

1. Patient with liver dysfunction
2. Patient with drug-resistant
3. Severe Malnutrition
4. Refuse to be involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Sputum Conversion Duration | six month after the intervention started
  Sputum conversion duration defined as the duration to change positive result in sputum smear into negative results. The sputum smear level using Ziehl Neelsen ranging from Negative to 3+.
Chest X-Ray Extension | Changes of number of active tuberculosis feature from baseline to 6 months
  Distribution of active tuberculosis feature in Chest X-Ray including number of consolidation and cavitation
Interleukin 6 Level | Changes of Interleukin 6 Level from baseline to 6 months
  Value of Interleukin 6 in blood Sample
Interleukin 10 Level | Changes of Interleukin 10 value from baseline to 6 months
  Value of Interleukin 10 in blood Sample

SECONDARY OUTCOMES:
Cluster Differentiation 4 (CD4) cells value | Changes of Cluster Differentiation 4 (CD4) cells value from baseline to 6 months
  Cluster Differentiation 4 (CD4) cells value in blood sample
Cluster Differentiation 8 (CD8) cells value | Changes of Cluster Differentiation 8 (CD8) cells value from baseline to 6 months
  Cluster Differentiation 8 (CD8) cells value in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Djamaludin Ma'dolangan, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Labuang Baji General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data including de-identified data and protocol

REFERENCES:
- [Background] Matar, C., Graham, E. 2017. Immune Modulatory Function. Clinician's Guide To AHCC, Evidence-Based Nutritional Immunotherapy, Edited by Anil D.K, Philip, C and Toshinori Ito. P.54-61.
- [Background] Suknikhom W, Lertkhachonsuk R, Manchana T. The Effects of Active Hexose Correlated Compound (AHCC) on Levels of CD4+ and CD8+ in Patients with Epithelial Ovarian Cancer or Peritoneal Cancer Receiving Platinum Based Chemotherapy. Asian Pac J Cancer Prev. 2017 Mar 1;18(3):633-638. doi: 10.22034/APJCP.2017.18.3.633. PMID 28440968
- [Background] Sun B, Wakame K, Sato E, Nishioka H, Aruoma OI, Fujii H. The effect of active hexose correlated compound in modulating cytosine arabinoside-induced hair loss, and 6-mercaptopurine- and methotrexate-induced liver injury in rodents. Cancer Epidemiol. 2009 Oct;33(3-4):293-9. doi: 10.1016/j.canep.2009.07.006. Epub 2009 Aug 20. PMID 19699163
- [Background] Terakawa N, Matsui Y, Satoi S, Yanagimoto H, Takahashi K, Yamamoto T, Yamao J, Takai S, Kwon AH, Kamiyama Y. Immunological effect of active hexose correlated compound (AHCC) in healthy volunteers: a double-blind, placebo-controlled trial. Nutr Cancer. 2008;60(5):643-51. doi: 10.1080/01635580801993280. PMID 18791928